CLINICAL TRIAL: NCT06306547
Title: Clinical Study Cohort of Idiopathic Inflammatory Myositis
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Principal Investigator, Qiong Fu, Director, RenJi Hospital
Other Study IDs: IIM001
Record Dates: First submitted 2024-02-21; First posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-02

CONDITIONS: Idiopathic Inflammatory Myopathies
MeSH Terms: conditions — Myositis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IMM patients with tumors: Patients with IMM will be grouped according to the type of positive myositis-specifc autoantibody,and then again according to whether and what type of tumor they had comorbid.
  Interventions: Other: no interventions were involved
- IMM patients without tumors: Patients with IMM will be grouped according to the type of positive myositis-specifc autoantibody,and then again according to whether and what type of tumor they had comorbid.
  Interventions: Other: no interventions were involved

INTERVENTIONS:
Other: no interventions were involved — no interventions were involved

SUMMARY:
Idiopathic inflammatory myositis (IIM), also known as myositis, are a heterogeneous group of diseases characterized by chronic inflammation of striated muscles and skin, with different clinical manifestations, treatment responses, and prognosis. This project will build a clinical follow-up cohort for idiopathic inflammatory myositis (IIM) centered on Renji Hospital, Shanghai Jiao Tong University School of Medicine, to promote the clinical and pathogenesis of this group of diseases.

ELIGIBILITY:
Inclusion Criteria:Subjects must meet the following criteria for inclusion in this study: meet the 2017 EULAR/ACR classification criteria for inflammatory myopathy (IIM) or the 2018 ENMC-DM classification criteria (see above), plus:

1. Age≥ 18 years old and ≤ 75 years old
2. Meet the 2017 EULAR/ACR classification criteria for inflammatory myopathy (IIM), the above score ≥ 5.5 points if there is no muscle biopsy, and 6.7 points ≥ if there is muscle biopsy
3. Cooperate with follow-up, examination and treatment and voluntarily sign the informed consent form.

   -

   Exclusion Criteria:Potential subjects who meet the inclusion criteria will be excluded if they meet any of the following criteria:

   a. IIM with other connective tissue diseases; b. Negative myositis antibody test; c. Those who are in the period of acute infection, or have a history of active tuberculosis in the past; d. People with allergies or allergies to multiple drugs; e. Those who have mental illness or other reasons and cannot cooperate with examination, follow-up or treatment; f. Women who are pregnant, or are trying to become pregnant; g. Those who are participating in or have participated in clinical trials within the specified time.

   -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aged 18-75 years and eligible for the 2017 European League Against Rheumatism/American College of Rheumatology.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2034-04-01 (Estimated); Study Completion 2034-04-01 (Estimated)

PRIMARY OUTCOMES:
High Resolution Computed Tomography of Chest | three months
  High Resolution Computed Tomography of Chest will be used to assess the incidence of interstitial pneumonia.
Cutaneous Disease Area and Severity Index | three months
  Cutaneous Disease Area and Severity Index will be used to assess the the severity of the rash.
Forced vital capacity | three months
  t refers to the maximum amount of air that cr trying to inhale as quickly as possible.
Manual Muscle Testing | three months
  Manual Muscle Testing will be used to assess patients with muscle weakness.
Forced expiratory volume in one second | three months
  It refers to the volume of the maximum exhalation exhaled in the first second of the maximum deep inhalation.

SECONDARY OUTCOMES:
Serum creatine kinase | three months
  Serum creatine kinase will be used to assess the disease activity in idiopathic inflammatory myopathies.